CLINICAL TRIAL: NCT04887428
Title: Occupational Insertion and Educational Level of Adult Patients With Pediatric Early Inflammatory Bowel Disease (IBD)
Acronym: PROMICI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017_19; 2017-A03397-46 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this project is to assess the occupational insertion of these adult patients with pediatric-onset IBD and to compare it with the general population.

The secondary objectives are:

1. to assess the level of education and compare it to that of the general population
2. to assess occupational insertion and the educational level according to:

   * The disease (Crohn's disease, ulcerative colitis or unclassified colitis)
   * sex
   * Age at diagnosis (<or ≥ 10 years)
   * The occurence of surgery, the location of the disease, the treatments undertaken
   * Quality of life
3. Evaluate the patient's feelings about the impact of his illness on occupational insertion and the educational level
4. To describe the quality of life of patients in relation to disease activity and health states (QALY calculation)
5. To assess the responsivness to change of the functional handicap score IBD-DI (n = 200 patients)

DETAILED DESCRIPTION:
Chronic inflammatory bowel diseases (IBD) are responsible for high morbidity and impaired quality of life of patients throughout disease course.

Numerous studies have shown the impact of the disease on the quality of life of patients with IBD. However, very little data is available on the level of education and professional integration of patients who started their IBD in childhood.

The hypothesis behind the study project is that the level of education and consequently the professional integration of patients with early pediatric IBD: 1) could be different from those of the general population; 2) and that these differences could be influenced by the nature of IBD, the age of its onset and its main characteristics.

The main objective of this project is to assess the professional integration of these adult patients with pediatric-onset IBD and to compare it with the general population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 25 and over at the time of the study
* Subject listed in the EPIMAD registry suffering from certain or probable Crohn's disease, or certain or probable ulcerative colitis, or certain or probable ulcerated proctitis, unclassified colitis, diagnosed between 01/01 / 1988 and 12/31/2011, with an age at diagnosis of less than 17 years (definition of the pediatric cohort of the EPIMAD Registry)
* Patient residing in the area of the EPIMAD registry: Nord, Pas-de-Calais, Somme or Seine-Maritime
* Patient not opposed to the research
* Patient not having objected to the use of their data for ancillary studies when registering in the EPIMAD register

Exclusion Criteria:

* None

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pediatric-onset IBD (diagnosed before the age of 17) and aged over 25 at the time of the study.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2019-11-28 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Rate of active workers in employment | through study completion, an average of 18 months
  Rate of active workers in employment collected using a standardized self-questionnaire

SECONDARY OUTCOMES:
Educational level | through study completion, an average of 18 months
  Description of educational level collected using a standardized self-administered questionnaire
Association between occupational insertion and disease variables | through study completion, an average of 18 months
  Associated factors are : disease type (Crohn / Ulcerative colitis), gender, location of the disease at diagnosis, surgery, treatments, age at diagnosis
Association between occupational insertion and quality of life | through study completion, an average of 18 months
  Quality of life as measured by SIBDQ questionnaire.
Association between educational level and disease variables | through study completion, an average of 18 months
  Associated factors are : disease type (Crohn / Ulcerative colitis), gender, location of the disease at diagnosis, surgery, treatments, age at diagnosis
Association between educational level and quality of life | through study completion, an average of 18 months
  Quality of life as measured by SIBDQ questionnaire.
Percentage of patients for whom the disease had an influence on the choice of studies | through study completion, an average of 18 months
  This question is directly asked to the patient and reflects its own feeling
Percentage of patients for whom the disease had an influence on the course of the studies | through study completion, an average of 18 months
  This question is directly asked to the patient and reflects its own feeling
Percentage of patients for whom the disease had an influence on the choice of profession | through study completion, an average of 18 months
  This question is directly asked to the patient and reflects its own feeling
Quality of life as measured by EQ5D-5L questionnaire | through study completion, an average of 18 months
  Quality of life as measured by EQ5D-5L questionnaire and transformed into utility according to French reference values. Quality of life will be described according to age, disease activity and surgery.
Disease activity for Crohn's patients | through study completion, an average of 18 months
  As measured by HBI (Harvey-Bradshaw Index). Disease activity will be used to describe quality of life according to disease state and to assessed sensitivity to change of IBD-Disability Index.
Disease activity for Ulcerative Colitis patients | through study completion, an average of 18 months
  As measured by SCCAI questionnaire (Simple Clinical Colitis Activity Index). Disease activity will be used to describe quality of life according to disease state and to assessed sensitivity to change of IBD-Disability Index.
Disability in 200 patients | through study completion, an average of 18 months
  As measured by IBD-DI (IBD Disability Index) in 200 patients previously questioned in 2012 in order to address the question of sensitivity to change of IBD-DI. Measure of change is disease activity as measured by HBI-Index for Crohn's patients and SCCAI for Ulcerative Colitis patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Turck, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Jeanne de Flandre Chu Lille, Lille, France